CLINICAL TRIAL: NCT05890066
Title: Effectiveness and Safety of Single-port Versus Multi-port Laparoscopic Surgery in the Treatment of Ectopic Pregnancy
Brief Title: Single-port Versus Multi-port Laparoscopic Surgery for Ectopic Pregnancy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hung Vuong Hospital (Other)
Responsible Party: Principal Investigator, Tri Bao Nguyen, Principle investigator, Hung Vuong Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 5863
Record Dates: First submitted 2023-05-25; First posted 2023-06-06 (Actual); Last update posted 2023-06-07 (Actual); Status verified 2023-06

CONDITIONS: Ectopic Pregnancy
Keywords: Laparoscopic surgery; Single-port laparoscope; Multi-port laparoscope
MeSH Terms: conditions — Pregnancy, Ectopic

STUDY DESIGN:
Intervention Model Description: The study is a parallel-group randomized control trial with 2 arms. Arm 1 includes patients who will be treated by traditional multi-port laparoscopic surgery. Aim 2 includes patients who will be treated by single-port laparoscopic surgery. All patients are randomized using computer-generated sequences with allocation ratio 1:1. This is a non-blinded study where all patients and surgical teams know the treatment option.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 4-port laparoscopic surgery (No Intervention): Patients with ectopic pregnancy will receive 4-Port laparoscopic surgery
- 1-port laparoscopic surgery (Experimental): Patients with ectopic pregnancy will receive 1-port laparoscopic surgery
  Interventions: Procedure: single-port laparoscopy

INTERVENTIONS:
Procedure: single-port laparoscopy — Compare the effectiveness and safety between single-port and multi-port laparoscopic surgery
  Arms: 1-port laparoscopic surgery

SUMMARY:
This study aims to compare the effectiveness and Safety of Single-port Versus Multi-port Laparoscopic Surgery in the Treatment of Ectopic Pregnancy

DETAILED DESCRIPTION:
Single-port laparoscopic surgery has become one of the treatment options for ectopic pregnancy with certain advantages such as reduced numbers of incision and scars, and increased patient's satisfaction post-surgery. At Hung Vuong hospital, the investigators do not have data about the application potential of single-port laparoscopic surgery for ectopic pregnancy treatment. Therefore, the investigators carry out this project to compare the effectiveness and safety of single-port versus traditional multi-port laparoscopic surgery in the treatment of ectopic pregnancy.

ELIGIBILITY:
Inclusion Criteria:

* 18 years old or older pregnant women who are indicated for laparoscopic surgery in the treatment of ectopic pregnancy.
* Agree to participate and give a consent

Exclusion Criteria:

* Allergic reactions to anesthetics
* Hemodynamic instability
* Ruptured ectopic pregnancy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — The investigators only recruit patients with ectopic pregnancy to participate in the study
Enrollment: 100 (Estimated)
Dates: Start 2023-11-01 (Estimated); Primary Completion 2024-05-31 (Estimated); Study Completion 2024-05-31 (Estimated)

PRIMARY OUTCOMES:
Blood loss | Immediately post surgery
  Measure the amount of blood loss
Surgical time | Immediately post surgery
  How long will it take for single-port vs multi-port surgical procedures

SECONDARY OUTCOMES:
Pain intensity | Within 4 weeks post surgery
  Use visual analogue scale to measure
Surgical complications | Within 4 weeks post surgery
  Organ damages, surgical site infections, pneumoperitoneum
Hospital stay | Within 4 weeks post surgery
  How long will be the recovery time

CONTACTS AND LOCATIONS:
Overall Officials: Nghiem X Huynh, Doctor, Study Director — Hung Vuong Hospital

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-04-28): https://cdn.clinicaltrials.gov/large-docs/66/NCT05890066/Prot_SAP_001.pdf